CLINICAL TRIAL: NCT01525693
Title: Evaluation of Effectiveness of Treatment Paradigm for Newly Diagnosed Type 2 Diabetes Patients in China (NEW2D STUDY) A Study Of China Cardiometabolic Registries (CCMR)
Brief Title: Evaluation of Effectiveness of Treatment Paradigm for Newly Diagnosed Type 2 Diabetes Patients in China
Acronym: NEW2D
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China Cardiometabolic Registries (Network)
Collaborators: Bristol-Myers Squibb (Industry); VitalStrategic Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CCMR--304-NEW2D
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; diabetics; high glucose; Chinese patients
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnosed within 6 months: No (test) intervention to be adminisitered

SUMMARY:
This is a study to gain better understanding on how those patients who are newly diagnosed with type 2 diabetes are treated and monitored. The study will record information such as type of therapy, therapeutic outcomes, and patients' satisfaction.

DETAILED DESCRIPTION:
The prevalence of diabetes around the world has increased from 30 million in 1985 to the current 235 million, and is expected to grow to 300 million in 2030, with more than 75 percent occurring in countries such as India and China. In China, economic prosperity and changes in diet and lifestyles have resulted in steep increase in prevalence of overweight, obesity, and diabetes. According to the latest study, in adults of 20 years of age or older, the incidence of diabetes has reached 9.7% and the prevalence 92.4 million. In a nationwide, cross over cohort study that was recently completed in China, the results showed that the duration of diabetes is positively correlated with the incidence of CAD and all microvascular diabetic complications. Preventing diabetes progression and preventing the onset of cardiovascular diseases early on at the stage of newly diagnosis is thus one of the most important goals in managing type 2 diabetes.

According to the Chinese Guidelines for Prevention and Treatment of Diabetes, which is consistent with IDF Clinical Guidelines Task Force Global Guideline for Type 2 Diabetes, the therapeutic target for type 2 diabetes is defined as HbA1C < 6.5%. Various national surveys conducted in China in 2003, 2004, 2006 have shown that only about one forth of type 2 diabetes patients in China reached this therapeutic target.Over the recent few years, a number of new antidiabetic treatments, such as DPP-IV inhibitors, have been introduced to the real world practice of diabetes management in China, creating exciting opportunities to potentially improve glycemic control. UKPDS (United Kingdom Prospective Diabetes Study) provided the evidence for improving glycemic control through aggressive treatment in western population. There is now substantial evidence on management of patients with type 2 diabetes. However, it is believed that not all patients have benefited from optimal diabetes management in China, partially due to diversity of standards of clinical practices and complexity of diabetes care itself. For example, it is unclear which treatment regimen works more effectively for managing newly diagnosed type 2 diabetes patients or whether a more aggressive strategy be used during the early stage of treatment. Moreover, it remains answering that what other factors may influence the treatment outcomes. There are clearly significant unmet needs and thus significant opportunities to leverage the existing medical advancement.

This study is thus designed to evaluate current treatment patterns and treatment outcomes for managing newly diagnosed type 2 diabetes patients and to assess specific unmet needs, influencing factors, management platforms, and gaps and trends in practice, providing a comprehensive knowledge in current management of newly diagnosed diabetes and insight on opportunities and strategy for future research and development of improved therapy.

ELIGIBILITY:
* 20 years of age or older
* Confirmed diagnosis of type 2 diabetes made within past 6 months according to the 2010 Chinese Guideline for Type 2 diabetes
* Have not received any pharmacological treatment for T2D, or have started on one regimen and have not switched or added any other hypoglycemic agent
* Have completed a lab test +/- 30 days of the baseline visit or is due for a lab evaluation including HbA1C, serum glucose, lipid profile, and other routine tests
* Willing to return for all follow up visits.

Exclusion Criteria:

* Patients who are not willing or not able to return to the same hospital for follow up visits every 3 months for one year after enrollment (e.g. do no reside locally)
* Patients who are participating in another interventional clinical trials
* Patients who are not willing to sign informed consent form

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects seen at outpatient clinics of tier 1, 2, and 3 hospitals across the 6 major geographic regions
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-10 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of this study is the overall proportion of patients whose HbA1c is less than 6.5%, measured at the end of one year follow up. | 12 months

SECONDARY OUTCOMES:
The proportions of patients receiving various regimen, and the duration of each regimen | 12 months
The clinical effectiveness of each regimen measured by the proportion of patients reaching the target glycemic control | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, MD, Principal Investigator — Peking University People's Hospital
Locations (2):
- China (2):
  - People's Hospital of Peking University, Beijing
  - Xijing Hospital, Xi'an

REFERENCES:
- [Derived] Luo Y, Wu H, Liao X, Zhao T, Cui N, Li A, Sun X, Zhang P, Huang Y, Zhang X, Yin H, Ji L. A Guideline-Based Decision Tree Achieves Better Glucose Control with Less Hypoglycemia at 3 Months in Chinese Diabetic Patients. Diabetes Ther. 2021 Jul;12(7):1887-1899. doi: 10.1007/s13300-021-01075-1. Epub 2021 May 29. PMID 34050897
- [Derived] Cai X, Hu D, Pan C, Li G, Lu J, Ji Q, Su B, Tian H, Qu S, Weng J, Zhang D, Xu J, Ji L. The risk factors of glycemic control, blood pressure control, lipid control in Chinese patients with newly diagnosed type 2 diabetes _ A nationwide prospective cohort study. Sci Rep. 2019 May 22;9(1):7709. doi: 10.1038/s41598-019-44169-4. PMID 31118445
- See also: Related Info — http://www.ccmregistry.org